CLINICAL TRIAL: NCT07243769
Title: A Pilot Randomized Controlled Trial Comparing Core Exercise, Aerobic Exercise, and Combined Exercise in Patients Undergoing Phase II Cardiac Rehabilitation.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202507175RINC
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Clinically Stable Myocardial Infarction or Heart Failure Patients; Heart Failure; Myocardial Infarction (MI)
MeSH Terms: conditions — Heart Failure; Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Core Exercise group (Experimental): tow sessions core exercise training per week
  Interventions: Other: Core exercise training
- Aerobic exercise group (Active Comparator): two sessions aerobic training per week
  Interventions: Other: conventional cardiac rehabilitation (aerobic training)
- Combined exercise group (Active Comparator): one session core exercise training and one session aerobic training per week
  Interventions: Other: combined training

INTERVENTIONS:
Other: Core exercise training — Two core sessions per week, 1 hour per session. Pilates-based core endurance training progressing in difficulty with emphasis on breathing and posture; exercises performed in sitting, supine, prone, and quadruped positions.
  Arms: Core Exercise group
Other: conventional cardiac rehabilitation (aerobic training) — Two aerobic training sessions per week, 1 hour per session. Aerobic program targets 40-80% heart-rate reserve on a treadmill or cycle ergometer.
  Arms: Aerobic exercise group
Other: combined training — One core training session and one aerobic training session per week, 1hr per session. Core program (Pilates-based) progresses in difficulty with emphasis on breathing and posture; aerobic program targets 40-80% heart-rate reserve on a treadmill or cycle ergometer.
  Arms: Combined exercise group

SUMMARY:
Cardiac rehabilitation (CR) is recommended after myocardial infarction (MI) or heart failure (HF), yet the added value of core muscle endurance training within CR remains uncertain. This randomized, three-arm trial will enroll 60 adults with stable MI or HF who are referred to Phase II CR. After consent and baseline testing, participants are allocated 1:1:1 to: (1) Pilates-based core endurance training, (2) standard aerobic CR (treadmill or cycle), or (3) combined aerobic plus core training. Supervised sessions occur twice weekly for eight weeks (~60 minutes/session) with continuous safety monitoring. The primary aim is to evaluate feasibility and safety of core training in this population. The study also compares effects of the three programs on cardiorespiratory fitness and function (e.g., peak oxygen uptake, six-minute walk distance), core endurance, balance, symptoms, and health-related quality of life. Findings will clarify whether adding core training improves outcomes and inform clinical exercise prescription in CR.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Diagnosed with myocardial infarction or heart failure with stable condition, and referred for participation in Phase II cardiac rehabilitation.
* Able to regularly attend training sessions twice a week.

Exclusion Criteria:

* Underwent cardiac surgery within the past three months.
* Presence of a pacemaker, defibrillator, or left ventricular assist device.
* Cognitive impairment or dementia that prevents understanding or following training instructions.
* Inability to complete cardiopulmonary exercise testing.
* Pregnancy.
* Contraindications to cardiac rehabilitation based on the American College of Sports Medicine (ACSM) guidelines, such as unstable angina, uncontrolled severe hypertension (resting systolic BP >180 mmHg or diastolic BP >110 mmHg), orthostatic hypotension (drop in BP >20 mmHg upon position change), severe aortic stenosis, uncontrolled severe arrhythmia, decompensated heart failure, third-degree atrioventricular block, acute pericarditis or myocarditis, aortic dissection, acute pulmonary embolism, or other acute medical conditions such as infection or fever.
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen uptake | Week 0 and after 8-week training program
  The peak oxygen uptake (VO₂peak) is measured using a cardiopulmonary exercise testing (CPET).

SECONDARY OUTCOMES:
Six-minute walk distance | Week 0 and after 8-week training program
  Participants are instructed to walk back and forth as quickly as possible along a flat, hard-surfaced indoor corridor for six minutes. The total distance walked within six minutes is recorded.
One-leg stand test | At Week 0 and after 8-week training program
  Participants stand barefoot on one leg, keeping the opposite leg lifted without touching the supporting leg. Hands are placed on the hips, and eyes are open, gazing forward. The maximum duration of stable standing is recorded. Each leg is tested twice, and the best score is used for analysis.
Plank endurance | At Week 0 and after 8-week training program
  Participants assume a forearm plank position, maintaining a straight trunk with core engaged. The duration for which the position is held is recorded. The body must remain in a straight line from head to heels, with no sagging of the hips.
Side plank endurance | At Week 0 and after 8-week training program
  Participants perform side planks on the left and right sides, supporting the body with one forearm while keeping the body in a straight line. The holding time for each side is recorded separately.
Trunk flexor endurance test | At Week 0 and after 8-week training program
  Performed using McGill's trunk flexor endurance protocol. Participants sit on a 60-degree inclined board with hips and knees bent at 90 degrees and arms crossed over the chest. The support board is then removed, and participants are asked to maintain the trunk at a 60-degree angle from the ground for as long as possible. The test ends when the participant can no longer hold the position.
Lumbo-pelvic control test | At Week 0 and after 8-week training program
  Participants lie supine in a crook-lying position (knees bent) with a pressure biofeedback unit placed under the third lumbar vertebra, inflated to 40 mmHg. Participants are instructed to slowly lift both legs to 90° hip flexion. If the pressure change is less than 10 mmHg during lifting, it is considered a success, indicating stable lumbar control; a change greater than 10 mmHg indicates failure due to uncontrolled lumbar flexion. Participants then lower both legs from 90° to 45° hip flexion. If the pressure change is less than 10 mmHg, it is considered a success, indicating good lumbar stability; a change greater than 10 mmHg indicates failure due to uncontrolled lumbar extension.
30 seconds sit to stand test | From enrollment to the end of treatment at 8 weeks
  Participants sit on an armless chair with arms crossed over the chest and are instructed to stand up and sit down as many times as possible within 30 seconds. The total number of full sit-to-stand repetitions is recorded.
Hand grip strength | From enrollment to the end of treatment at 8 weeks
  Participants sit with the dominant arm relaxed at the side, elbow flexed at 90°, and hold a hand dynamometer. They are instructed to squeeze maximally for 2-3 seconds. Three trials are performed with 30-second rest intervals, and the highest value is recorded as the maximal handgrip strength.
Time to exhaustion at 80% of VO₂peak | At Week 0 and after 8-week training program
  Based on the results of the baseline cardiopulmonary exercise test, participants perform a constant-load exercise at 80% of their VO₂peak until volitional exhaustion or until reaching test termination criteria. The total exercise time to exhaustion is recorded.
Body composition | At Week 0 and after 8-week training program
  Body fat percentage and lean body mass are measured using bioelectrical impedance analysis (BIA).

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No